CLINICAL TRIAL: NCT02603471
Title: Cell Phone Technology Targeting ART and Naltrexone Adherence and Alcohol Use
Acronym: ALCTXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Suzette Glasner-Edwards, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALCTEXT
Record Dates: First submitted 2014-07-15; First posted 2015-11-11 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: HIV Infections; Alcohol Dependence
Keywords: HIV infections; Alcohol dependence; Mobile Technology
MeSH Terms: conditions — HIV Infections; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Text Messaging CBT (TXT-CBT) (Experimental): This condition will receive CBT based text messaging (TXT-CBT). Those assigned to TXT-CBT will also be given a treatment manual (developed in Phase I) containing descriptions of core therapeutic content/topics for each week. HIV-infected participants will have an initial meeting with a CBT clinician to review the Life-Steps concepts. The 3 most applicable medication adherence skills will be identified for emphasis in tailored messages. A research coordinator will meet with the participants weekly at data collection visits throughout the intervention phase to answer any technical questions and ensure that the intervention program is working properly.
  Interventions: Behavioral: Text Messaging CBT (TXT-CBT)
- Informational group (Active Comparator): A pamphlet with information about HIV, the importance of ART adherence, and relapse prevention will be provided to participants in this condition.
  Interventions: Other: Informational group

INTERVENTIONS:
Other: Informational group — A pamphlet will be provided to the participants with information about ART adherence, HIV and relapse prevention.
  Arms: Informational group
Behavioral: Text Messaging CBT (TXT-CBT) — Those assigned to TXT-CBT will be given a treatment manual (developed in Phase I) containing descriptions of core therapeutic content/topics for each week. HIV-infected participants will have initial meeting with a CBT clinician to review the core CBT concepts for promoting ART adherence. The 3 most applicable medication adherence skills will be identified for emphasis in tailored messages. A research coordinator will meet with the participants weekly at data collection visits throughout the intervention phase to answer any technical questions and ensure that the intervention program is working properly.
  Arms: Text Messaging CBT (TXT-CBT)

SUMMARY:
The proposed study, for HIV positive alcohol dependent adults currently taking naltrexone, is a pilot randomized controlled trial (RCT) examining the outcomes of a 12-week behavioral support program delivered via text-messaging.

It is expected that the text messaging intervention will reduce alcohol use and HIV-risk behaviors. The investigators also hypothesize that the intervention will improve adherence to HIV treatment and naltrexone.

To test the effects of the intervention on these target outcomes, 25 participants receiving the text messaging intervention will be compared to 25 participants receiving an informational pamphlet. The pamphlet will contain information about the importance of HIV treatment adherence, reducing HIV risk behaviors, and health consequences associated with alcohol use.

By providing support to maximize HIV treatment regimen and naltrexone adherence, coupled with coping skills to promote abstinence from alcohol, the text messaging intervention may provide a promising, cost-effective, and easily deployable behavioral support program for alcohol users who are HIV-infected.

DETAILED DESCRIPTION:
The aims of this study are to: 1) implement and evaluate a 12-week cognitive behavioral therapy (CBT) intervention using text messaging via mobile phone technology (ALC-TXT-CBT) to reduce alcohol use, reduce HIV-risk behaviors and facilitate medication adherence in a population of alcohol dependent adults with HIV-infection and 2) examine potential mechanisms of action of ALC-TXT-CBT. The investigators hypothesize that ALC-TXT-CBT will produce greater reductions in alcohol use and HIV-risk behaviors, and will improve HIV treatment regimen and naltrexone (Vivitrol) adherence, relative to the control condition (informational pamphlet).

Further, the investigators expect that ALC-TXT-CBT will facilitate greater changes in negative affect, self-efficacy, and social support, and these changes will be associated with substance use outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older;
2. DSM-IV diagnosis of Alcohol Dependence;
3. Use of 5 or more standard drinks per drinking day for men or 4 or more for women (over the past 30 days);
4. HIV-infected serostatus;
5. Able to provide informed consent;
6. Willing and able to participate in study procedures,
7. Good general health or, in the case of a medical/psychiatric condition needing ongoing treatment, potential participant should be under the care of a physician who provides documented willingness to continue participant's medical management and coordinate care with the study physicians.
8. Adherent to <90% of antiretroviral therapy regimen, as determined by the medication adherence screening procedure
9. Currently taking or interested in taking/receiving more information about naltrexone in its injectable form (Vivitrol). Participants WILL NOT be prescribed or given naltrexone as part of this study. Participants not currently on vivitrol will be referred to a physician in the community to be evaluated for vivitrol eligibility and to receive vivitrol if applicable.
10. Owning a cell phone. Participants are required to own their phone and cannot use someone else's phone.

Exclusion Criteria:

1. Presence of serious medical condition that would, in the opinion of the study physician, make participation medically hazardous (e.g., acute hepatitis, unstable cardiovascular, liver or renal disease).
2. A current pattern of alcohol or sedative use, as assessed by the study physician, which would preclude safe participation in the study and/or would likely require imminent medical detoxification.
3. Has undergone more than one inpatient medical detoxification treatment;
4. Lack of proficiency in English;
5. Currently homeless (unless residing in a recovery home for which contact information can be provided);
6. Presence of clinically significant psychiatric symptoms as assessed by MINI, such as psychosis, acute mania, or suicide risk that would require immediate treatment or make study compliance difficult.
7. Not currently taking naltrexone in its injectable form (Vivitrol) or not interested in taking/receiving information about vivitrol or not interested in taking vivitrol
8. Adherent to > or =90% of antiretroviral therapy regimen, as determined by the medication adherence screening procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change Outcome Measure: Substance Use (ASI) | baseline (week 0), treatment-end (week 12), and Follow-Up (FU) (week 24)
  Addiction Severity Index (ASI) is an instrument widely used in addiction research to quantify drug use frequency and related problem areas.
Change Outcome Measure: HIV Risk (RBRA) | RBRA will be collected at baseline (week 0), treatment-end (week 12), and FU (week 24)
  Risk Behavior Survey (RBRA): The RBRA is a brief interview assessing involvement in HIV risk behaviors in the areas of drug use and sex in the previous 30 days. Additional items include whether the sexual partner uses or injects drugs. The participants' change in RBRA scores is being assessed from each timepoint to the next.
Change Outcome Measure: Adherence Measures | Baseline, Weeks 4,8,12,16,20 and 24
  ART Adherence. The investigator will use monthly phone-based unannounced pill counts (UPCs).
Change Outcome Measure: Substance Use (UDS) | UDS is collected at baseline, week 4, week 8, week 12 and week 24
  Urine Drug Screen (UDS). Urine drug screens will be collected monthly using temperature controlled test cups. An FDA-approved one-step test will be used. During the 12-week treatment period, one full-screen panel and two panels only testing for opioids (heroin and prescription opioids) will be conducted. The UDS will test for the presence of: amphetamines, benzodiazepines, methadone, cocaine, methamphetamine, morphine (heroin), hydrocodone (Vicodin), oxycodone (OxyContin), and marijuana. The participants' change in substance use over time (as assessed by the ASI and UDS results) is being assessed from each timepoint to the next.
Change Outcome Measure: Viral Load | at baseline (week 0), treatment end (week 12), and FU (week 24).
  Viral load will serve as a biological indicator of adherence. Consistent with the typical frequency with which viral load is assessed in clinical settings, data concerning viral load will be collected at baseline (week 0), treatment end (week 12), and FU (week 24) via chart review from the participant's medical provider.

SECONDARY OUTCOMES:
Change in Quality of Life | Weeks 0,12 and 24
  Data concerning health-related quality of life during and after treatment will be collected using the SF-12 Health Survey. It measures eight health domains, and each survey provides psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Glasner, PhD, Principal Investigator — UCLA Integrated Substance Abuse Programs
Locations (1):
- UCLA Integrated Substance Abuse Programs, Los Angeles, California, United States

REFERENCES:
- [Derived] Glasner S, Chokron Garneau H, Ang A, Ray L, Venegas A, Rawson R, Kalichman S. Preliminary Efficacy of a Cognitive Behavioral Therapy Text Messaging Intervention Targeting Alcohol Use and Antiretroviral Therapy Adherence: A Randomized Clinical Trial. PLoS One. 2020 Mar 12;15(3):e0229557. doi: 10.1371/journal.pone.0229557. eCollection 2020. PMID 32163431